CLINICAL TRIAL: NCT03551288
Title: A Phase I, Single-Center, Single Dose Study to Evaluate the Effect of Food, Gender, and Age on Safety and Pharmacokinetic Profiles of SUVN-911 Tablets Orally Administered in Healthy Subjects
Brief Title: Effect of Food, Gender, and Age on the Pharmacokinetic Profile of SUVN-911 in Healthy Subjects
Acronym: SUVN-911
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP1S2911A4B2
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
Keywords: SUVN-911; Depression; alpha4 beta2 receptor
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in 1 of 3 cohorts; Cohort 1 (Food Effect Cohort), Cohort 2 (Gender Effect Cohort), and Cohort 3 (Age Effect Cohort). Subjects in Cohort 1 will receive a single oral dose of SUVN-911 on Day 1 under fasted or fed conditions and again on Day 8 under fasted or fed conditions (crossover design). Subjects in Cohort 2 and Cohort 3 will receive a single oral dose of SUVN-911 on Day 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Food Effect Cohort (Experimental): Twelve healthy male subjects 18 to 45 years of age, inclusive, will be administered a single oral dose of SUVN-911 on Day 1 (Period 1) and Day 8 (Period 2) with and without food in a crossover manner.
  Interventions: Drug: SUVN-911
- Gender Effect Cohort (Experimental): Eight healthy female subjects 18 to 45 years of age, inclusive, will be administered a single dose of SUVN-911.
  Interventions: Drug: SUVN-911
- Age Effect Cohort (Experimental): Eight healthy male subjects ≥ 65 years of age will be administered a single oral dose of SUVN-911.
  Interventions: Drug: SUVN-911

INTERVENTIONS:
Drug: SUVN-911 — Tablet

SUMMARY:
The purpose of the study is to investigate the effect of Food, Gender, and Age on the Pharmacokinetic Profile of SUVN-911 in Healthy Subjects

DETAILED DESCRIPTION:
This is a Phase I, single-center, open-label, single dose study to evaluate the effect of food, gender, and age on the safety and Pharmacokinetic profiles of single doses of SUVN-911, administered orally in healthy subjects.

The primary objective is to evaluate the effect of food, gender, and age on the pharmacokinetics of a single dose of SUVN-911 administered orally to healthy subjects.

The secondary objective is to evaluate the safety and tolerability of a single dose of SUVN-911 administered orally to healthy adult male, female, and elderly subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects, 18 to 45 years of age (inclusive) for Cohort 1, healthy female subjects, 18 to 45 years of age (inclusive) for Cohort 2, and healthy male subjects ≥ 65 years of age (inclusive) for Cohort 3, at the time of signing the informed consent.

Subjects in Cohorts 1 and 2 must have a body weight of at least 50 kg and body mass index (BMI) within the range of 18 to 30 kg/m2 (inclusive). Elderly subjects in Cohort 3 must have a body weight of at least 50 kg and BMI within the range of 18 to 32 kg/m2 (inclusive)

Exclusion Criteria:

History of any important clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.

History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.

Any clinically important illness, medical/surgical procedure, or trauma within 28 days of the first administration of the study treatment (Day 1).

Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.

Any positive result at Screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Area under concentration (AUC) | 24 hours
  Plasma concentration versus time

SECONDARY OUTCOMES:
Vital signs | 24 hours
  blood pressure determination

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lomeli, MD, Principal Investigator — IQVIA Phase One Services, LLC
Locations (1):
- IQVIA Phase One Services, LLC, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nirogi R, Benade V, Goyal VK, Pandey SK, Mohammed AR, Shinde A, Dogiparti D, Ravula J, Jetta S, Palacharla VRC. Safety, Tolerability, and Pharmacokinetics of Ropanicant (SUVN-911), a Novel Alpha4 Beta2 Nicotinic Acetylcholine Receptor (alpha4beta2 nAChR) Antagonist, in Healthy Adult and Elderly Subjects. Clin Drug Investig. 2022 Sep;42(9):747-762. doi: 10.1007/s40261-022-01189-9. Epub 2022 Aug 13. PMID 35963959